CLINICAL TRIAL: NCT04098562
Title: The Efficacy of LL-37 Cream on Aerobic Bacteria Colonization Pattern, Inflammation Response: Interleukin 1α (IL-1α) and Tumor Necrosis Factor α (TNF-α), and Healing Rate of Diabetic Foot Ulcers
Brief Title: Efficacy of LL-37 Cream on Bacteria Colonization, Inflammation Response and Healing Rate of Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Eliza Miranda, MD, Staff of Tropical Infection Division, Department of Dermatology and Venereology, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-09-1128
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): 0.5 mg/mL LL-37 cream, administered twice a week for 4 weeks
  Interventions: Drug: LL37; Procedure: Standard Wound Care
- Placebo (Placebo Comparator): Placebo cream, administered twice a week for 4 weeks
  Interventions: Procedure: Standard Wound Care

INTERVENTIONS:
Drug: LL37 — cream
  Arms: Treatment
Procedure: Standard Wound Care — Standard wound debridement

SUMMARY:
Diabetic foot ulcer (DFU) is a common complication of diabetes with global prevalence of 6.3%. Treatment of diabetic foot ulcer (DFU) is challenging with disappointing outcome. Wound debridement, infection control, pressure relief and revascularization are main pillars of DFU management. Various substances and modalities are being investigated for their potential effects in treating DFU, one of which is LL-37.

In this randomized, controlled trial, 40 patients with uncomplicated DFU will be enrolled. Patients are randomly assigned to undergo twice a week treatment with 0.5 mg/mL LL-37 cream (treatment group) or placebo cream (control group) for 4 weeks in addition to standard wound care. The primary outcomes are the healing rate measured by wound area and granulation index and changes in patterns of aerobic bacteria colonization during the 4-week study duration and changes in concentrations of IL-α and TNF-α from fluid collected from DFU on the end of the second and third week of study compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients with DFU
* Ankle brachial index (ABI) 0.9 - 1.3
* Wound area 5 - 20 cm^2
* Wound depth until subcutaneous tissue
* Without systemic infection, osteomyelitis, septic arthritis, or fasciitis
* Subjects are willing to participate by signing consent

Exclusion Criteria:

* Gangrene
* On treatment with systemic corticosteroids within 7 days before the start of study
* On treatment with systemic antibiotics within 2 days before the start of study
* Patients with end stage renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Healing Rate at 1 Week | Changes from baseline of granulation index at 1 week
  Measured by difference of granulation index by ImageJ
Changes of Healing Rate at 2 Week | Changes from baseline of granulation index at 2 weeks
  Measured by difference of granulation index by ImageJ
Changes of Healing Rate at 3 Week | Changes from baseline of granulation index at 3 weeks
  Measured by difference of granulation index by ImageJ
Changes of Healing Rate at 4 Week | Changes from baseline of granulation index at 4 weeks
  Measured by difference of granulation index by ImageJ
Changes of Aerobic Bacteria Count and Type of Bacteria Species at 1 Week | Changes from baseline of the species of bacteria grown on culture and the quantities of their colonies in CFU/swab at 1 week
  Measured by the species of bacteria grown on culture and the quantities of their colonies in CFU/swab
Changes of Aerobic Bacteria Count and Type of Bacteria Species at 2 Week | Changes from baseline of the species of bacteria grown on culture and the quantities of their colonies in CFU/swab at 2 week
  Measured by the species of bacteria grown on culture and the quantities of their colonies in CFU/swab
Changes of Aerobic Bacteria Count and Type of Bacteria Species at 3 Week | Changes from baseline of the species of bacteria grown on culture and the quantities of their colonies in CFU/swab at 3 week
  Measured by the species of bacteria grown on culture and the quantities of their colonies in CFU/swab
Changes of Aerobic Bacteria Count and Type of Bacteria Species at 4 Week | Changes from baseline of the species of bacteria grown on culture and the quantities of their colonies in CFU/swab at 4 week
  Measured by the species of bacteria grown on culture and the quantities of their colonies in CFU/swab
Changes of Inflammation Marker at 2 Week | Changes from baseline at the end of second week
  Measured by the concentrations of IL-α and TNF-α by ELISA
Changes of Inflammation Marker at 3 Week | Changes from baseline at the end of third week
  Measured by the concentrations of IL-α and TNF-α by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Eliza Miranda, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (3):
- Indonesia (3):
  - RS Persahabatan, Jakarta, DKI Jakarta
  - RS Pusat Angkatan Darat Gatot Soebroto, Jakarta Pusat, DKI Jakarta
  - RSUPN dr. Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miranda E, Bramono K, Yunir E, Reksodiputro MH, Suwarsa O, Rengganis I, Harahap AR, Subekti D, Suwarto S, Hayun H, Bardosono S, Baskoro JC. Efficacy of LL-37 cream in enhancing healing of diabetic foot ulcer: a randomized double-blind controlled trial. Arch Dermatol Res. 2023 Nov;315(9):2623-2633. doi: 10.1007/s00403-023-02657-8. Epub 2023 Jul 22. PMID 37480520